CLINICAL TRIAL: NCT01547104
Title: Effect of Linagliptin in Comparison With Glimepiride as Add on to Metformin on Postprandial Beta Cell Function, Postprandial Metabolism and Oxidative Stress in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marcus Borchert (Industry)
Collaborators: ikfe-CRO GmbH (Industry); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Marcus Borchert, Prof. Dr. Thomas Forst, ikfe-CRO GmbH
Organization: ikfe-CRO GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ikfe-Lina-002; 2012-000179-17 (EudraCT Number)
Record Dates: First submitted 2012-02-21; First posted 2012-03-07 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glimepiride-ratiopharm (Active Comparator): Glimepiride (1-4mg) as add on therapy
  Interventions: Drug: Glimepiride
- Trajenta (Experimental): Linagliptin 5 mg as add on therapy
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Linagliptin — Linagliptin dosed 5 mg as add on therapy to an existing metformin therapy
  Arms: Trajenta
Drug: Glimepiride — Glimepiride 1-4mg (individually dosed) as add on therapy to an existing metformin therapy
  Other Names: Glimepirid-ratiopharm
  Arms: Glimepiride-ratiopharm

SUMMARY:
The goal of this mechanistic study is to investigate the effect of Linagliptin in comparison to Glimepiride as add on therapy on several parameters characterizing postprandial metabolism and oxidative stress in type 2 diabetic patients on stable control with metformin.

DETAILED DESCRIPTION:
The goal of this mechanistic study is to investigate the effect of Linagliptin in comparison to Glimepiride as add on therapy on several parameters characterizing postprandial metabolism and oxidative stress in type 2 diabetic patients on stable control with metformin.

This mechanistic phase IV study has a prospective, comparative, open, randomized, two arm and exploratory design. Overall 40 Patients will be randomized to two treatment arms both receiving Metformin at a maximally tolerated dose. In addition to that both treatment groups will receive either an individually titrated dose of Glimepiride or 5mg once daily of Linagliptin. Subsequent to a standardized meal, several parameters reflecting beta cell function, metabolism and oxidative stress will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus type 2
2. HbA1c > 6.5% - ≤ 8.5%
3. HbA1c > 7.0% - ≤ 8.5% for those patients with a significant cardiovascular history
4. Treatment with metformin at a maximum tolerated dose
5. Age 45 - 75 years (inclusively)
6. Patient consents that his/her family physician/diabetologist will be informed of trial participation.

Exclusion Criteria:

1. Pretreatment with PPAR gamma agonists within the last three months
2. History of type 1 diabetes
3. Uncontrolled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >90 mmHg)
4. Acute infections
5. Medical history of hypersensitivity to the study drugs or to drugs with similar chemical structures
6. History of severe or multiple allergies
7. Treatment with any other investigational drug within 3 months before trial entry.
8. Progressive fatal disease
9. History of drug or alcohol abuse in the past 2 years
10. State after kidney transplantation
11. Serum potassium > 5.5 mmol/L
12. Pregnancy or breast feeding
13. Sexually active woman of childbearing age not practicing a highly effective method of birth control as defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs, sexual abstinence or vasectomized partner.
14. Acute myocardial infarction, open heart surgery or cerebral event (stroke/TIA) within the previous 30 days
15. Any elective surgery during study participation
16. Have had more than one unexplained episode of severe hypoglycemia (defined as requiring assistance of another person due to disabling hypoglycemia) within 6 months prior to screening visit
17. History of pancreatitis
18. History of dehydration, pre-coma diabeticum or diabetic ketoacidosis
19. Acute or scheduled investigation with iodine containing radiopaque material
20. Uncontrolled unstable angina pectoris
21. History of pericarditis, myocarditis, endocarditis
22. Recent pulmonary embolism
23. Hemodynamic relevant aortic stenosis
24. Aortic aneurysm
25. Regular use of NSAID's (no acute use of NSAID within 48 hours before V2,V4,V5)
26. Lack of compliance or other similar reason that, according to investigator, precludes satisfactory participation in the study
27. History of respiratory, gastrointestinal, hepatic (ALAT and/or ASAT > 3 times the normal reference range), renal (Creatinine > 1.1 mg/dl in women and > 1.5 mg/dl in men ), neurological, psychiatric and/or hematological disease as judged by the investigator
28. Lactose intolerance
29. Intake of Coumarin or coumarin derived compounds such as phenprocoumon (Marcumar) or warfarin (Coumadin, Warfant)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Postprandial increase in intact Proinsulin levels (Peak, AUC) | 30, 60, 90, 120, 150, 180, 210, 240, 270 300 mins post test meal procedure, 3 times within 12 weeks treatment
Postprandial Proinsulin/Insulin Ratio | after 12 weeks treatment
Fasting intact Proinsulin levels | after 12 weeks treatment
Fasting Proinsulin/Insulin Ratio | after 12 weeks treatment
Fasting Blood Glucose | after 12 weeks treatment
Postprandial Blood Glucose Excursions (Peak; AUC) | 30, 60, 90, 120, 150, 180, 210, 240, 270 300 mins post test meal procedure, 3 times within 12 weeks treatment
Fasting Lipids | after 12 weeks treatment
Postprandial Lipids | after 12 weeks treatment
Fasting Erythrocyte Flexibility | after 12 weeks treatment
Postprandial Erythrocyte Flexibility | after 12 weeks treatment
Fasting GLP-1 levels | after 12 weeks treatment
Postprandial GLP-1 levels | after 12 weeks treatment
Fasting cGMP | after 12 weeks treatment
Postprandial cGMP | after 12 weeks treatment
Fasting Calcitonin | after 12 weeks treatment
Fasting PAI-1 levels | after 12 weeks treatment
Postprandial PAI-1 levels | after 12 weeks treatment
Fasting ADMA levels | after 12 weeks treatment
Postprandial ADMA levels | after 12 weeks treatment
Fasting Malonyldialdehyd | after 12 weeks treatment
fasting oxidatively modified nucleosides 8-oxodG and 8-oxoGuo | after 12 weeks treatment

SECONDARY OUTCOMES:
Hypoglycemic events | after 12 weeks treatment
Body Weight | after 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forst, MD, PhD, Principal Investigator — Ikfe GmbH
Locations (1):
- ikfe GmbH, Mainz, Rhineland-Palatinate, Germany